CLINICAL TRIAL: NCT02704741
Title: Clinical Study of the CO2RE Laser Device Performance for Vaginal Atrophy Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF19731
Record Dates: First submitted 2016-02-28; First posted 2016-03-10 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Vaginal Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all subjects (Experimental): Eligible subjects will undergo 3 treatments in 4±1 weeks interval on the Vagina (External/Vulva and Internal/Vagina) with the CO2RE device according to study protocol.
  Subject will return for to 5 follow-up (FU) visits: 1 week ± 2 days post first treatment visit and 1, 3, 6 and 12 months after last (third) treatment (± 2 weeks).
  Methodology described in protocol to evaluate efficacy of treatments will be carried out at each visit at the clinic.
  Interventions: Device: CO2RE

INTERVENTIONS:
Device: CO2RE — The CO2RE system device is intended for dermatological procedures requiring ablation, coagulation and resurfacing of soft tissue, including skin

SUMMARY:
The CO2RE laser system is a fractional CO2 laser that is FDA approved under a 510(k) K101321 for dermatologic procedures requiring ablation and coagulation of soft tissues, including the skin Eligible subjects will undergo 3 treatments in 4±1 weeks interval on the Vagina (External/Vulva and Internal/Vagina) with the CO2RE device according to study protocol.

Subject will return for to 5 follow-up (FU) visits: 1 week ± 2 days post first treatment visit and 1, 3, 6 and 12 months after last (third) treatment (± 2 weeks).

Methodology described in protocol to evaluate efficacy of treatments will be carried out at each visit at the clinic.

DETAILED DESCRIPTION:
This study is a Prospective clinical study to demonstrate the CO2RE laser device for safety and efficacy for Vaginal Atrophy.

Up to a total of 60 healthy candidates, seeking vaginal treatment from the participating investigator will be enrolled at a participating study site. Subjects will receive three (3) CO2RE treatments.

Each subject will be followed for additional 5 post treatment visits (FU visits) that will be conducted at:

* One week post first treatment - 1wk FU ± 2 days (Safety).
* 1 month post last treatment - 1m FU ± 2 weeks (efficacy & Safety).
* 3 months post last treatment - 3m FU ± 2 weeks (efficacy & Safety).
* 6 months post last treatment - 6m FU ± 2 weeks (efficacy & Safety).
* 12 months post last treatment - 12m FU ± 2 weeks (efficacy & Safety).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects seeking treatment of Vaginal Atrophy in the vagina area (External - vestibule and introitus; Internal - Vaginal canal)
2. Healthy female subjects age greater than or equal to 35 years of age who are post menopausal for at least one year, for any reason whether surgical , chemical or natural.
3. Absence of menstruation for at least 12 months
4. Not responding to or satisfied with previous local estrogen therapy
5. Desire to maintain sexual activity
6. Informed consent process completed and subject signed consent
7. Willing to receive the proposed CO2RE treatment and follow-up protocol
8. Post-menopausal or surgically sterilized.
9. Normal cell cytology (PAP smear)
10. Negative urinalysis and a normal vaginal canal (no evidence of dysplasia and occult or active infection)
11. The external vaginal area (vestibule and introitus) free of injuries and bleeding
12. Subject experienced sexual activity at least once a month

Exclusion Criteria:

1. Subject had surgery or any other procedure for Vaginal Tightening in the last 12 months
2. Use of hormone replacement therapy, either systemic or local within the last 6 months prior to study
3. Lubricants or any localized preparation in the 30 days prior to enrollment
4. Patient with history of herpes.
5. Acute or recurrent urinary tract infection (UTI) or genital infection (e.g. herpes, candida)
6. Active malignancy or history of malignancy in the past 5 years
7. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
8. Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), lupus, porphyria, or pertinent neurological disorders (i.e. any disease state that in the opinion of the Physician would interfere with the treatment, or healing process)
9. Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician discretion)
10. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications
11. Suffering from hormonal imbalance, whether related to thyroid, pituitary, or androgen
12. History of significant lymphatic drainage problems
13. History of cancer which required lymph node biopsy or dissection
14. Suffering from significant conditions in the treated areas or inflammatory conditions, including, but not limited to, open lacerations or abrasions of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
15. History of keloid scarring, abnormal wound healing and / or prone to bruising
16. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders
17. Use of isotretinoin (Accutane®) within 6 months of treatment or during the study
18. Subject on systemic corticosteroid therapy 6 months prior to and throughout the course of the study
19. Dysplastic nevi in the area to be treated
20. Participation in a study of another device or drug within 6 month prior to enrollment or during this study, if treatments of vagina were involved
21. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study
22. Prolapse staged >_ II, according to the pelvic organ prolapse quantification (ICS-POP-Q) system
23. Previously undergone pelvic reconstructive surgery

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Vulvovaginal Symptom Questionnaire | Baseline, 1 , 2 , 3, 5, 8, and 14 months
  Vulvovaginal Symptom Questionnaire will be used to evaluate improvement of vulvovaginal atrophy symptoms.

SECONDARY OUTCOMES:
Number of participants with adverse events | throughout study duration, day 0 up to 17 months
  Number, severity and duration of adverse events following CO2 treatment
Vaginal Health Index Improvement | Baseline, 1 , 2 , 3, 5, 8, and 14 months
  Evaluation of vaginal wall conditions such as pH, elasticity, bleeding signs, secretion type and consistency and hydration.
Change from Baseline in Female Sex Function Index | Baseline, 1 , 2 , 3, 5, 8, and 14 months
  Female Sex Function Index will be used to evaluate improvement of vulvovaginal atrophy symptoms
Satisfaction questionnaire | 2 weeks and 1 , 2 , 3, 5, 8, and 14 months
  A questionnaire will be used to evaluate satisfaction with treatment outcome
Visual analog score for pain | day 0, 4 weeks, 8 weeks
  Patients will complete a visual analog scale to report pain level associated with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Konika Patel Schallen, MD, Study Director — Syneron Candela
Locations (4):
- United States (4):
  - FamWell.MD, Jacksonville, Florida
  - 6400 Dutchmans Pkwy Ste 335 Louisville, KY 40205 US, Louisville, Kentucky
  - Syneron-Candela Institute for Excellence, Wayland, Massachusetts
  - Dermatology and Laser Surgery Center of New York, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salvatore S, Nappi RE, Parma M, Chionna R, Lagona F, Zerbinati N, Ferrero S, Origoni M, Candiani M, Leone Roberti Maggiore U. Sexual function after fractional microablative CO(2) laser in women with vulvovaginal atrophy. Climacteric. 2015 Apr;18(2):219-25. doi: 10.3109/13697137.2014.975197. Epub 2014 Dec 16. PMID 25333211
- [Derived] Alexiades MR. Fractional Co2 Laser Treatment of the Vulva and Vagina and the Effect of Postmenopausal Duration on Efficacy. Lasers Surg Med. 2021 Feb;53(2):185-198. doi: 10.1002/lsm.23247. Epub 2020 Apr 23. PMID 32329093